CLINICAL TRIAL: NCT07155824
Title: Innovative Plant Proteins Fibre and Physical Activity Solutions to Modulate Whole Body and Skeletal Muscle Protein Metabolism in Older Adults
Brief Title: Impact of Plant Proteins and Exercise on Protein Metabolism in Older Adults
Acronym: APPETITE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Clermont-Ferrand (Other)
Collaborators: Institut National de Recherche pour l'Agriculture, l'Alimentation et l'Environnement (Other); Université d'Auvergne (Other); Friedrich-Alexander-Universität Erlangen-Nürnberg (Other); University College Dublin (Other); University of Padova (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: RBHP 2023 RICHARD 2; ANSM (Other: 2023-A01655-40)
Record Dates: First submitted 2024-07-22; First posted 2025-09-04 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-08

CONDITIONS: Eldery People; Sedentarity
MeSH Terms: interventions — Whey; Exercise

STUDY DESIGN:
Intervention Model Description: Controled, monocentric, open label study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Dietary proteins and physical activity (Experimental): Effect of physical activity program on protein metabolism following ingestion of whey or plant protein blend
  Interventions: Dietary Supplement: Whey and plant protein blend

INTERVENTIONS:
Dietary Supplement: Whey and plant protein blend — The 12 week intervention will involve 2 weekly group exercise sessions incorporating strength and balance exercises, along with home-based exercise focused on increasing time spent walking.
  Other Names: Physical activity

SUMMARY:
To gain mechanistic insights by examining the impact of innovative plant-protein fibre products, physical activity interventions on digestibility, amino acid bioavailability and whole-body protein metabolism in older persons

DETAILED DESCRIPTION:
Objective : to examine splanchnic extraction (SE), peripheral amino acid (AA) bioavailability and utilization (protein retention) from innovative plant proteins products, and muscle signalling markers before and after a physical activity (PA) program in inactive older persons

A randomized, crossover study including 12 inactive older men (65+ yrs) will be performed in order to compare the selected plant protein product to whey protein when included into a complete meal. During a kinetic day, each participant will consume alternatively, on 2 separate occasions, a test meal containing a plant protein mixture or 30 g whey protein. The methodology of stable isotope tracers: [15N] Leucine added to test meal and [1-13C] leucine administered intravenously will be used throughout a kinetic day, to evaluate the splanchnic extraction, the dietary amino acid bioavailability, and the whole body protein metabolism (protein synthesis, protein breakdown, AA oxidation and net balance). Carbon dioxide production rates will be measured by open-circuit indirect calorimetry. All measurements will be performed before the meal and post-prandial in regular intervals for 420 min.

In addition, postprandial plasma insulin and glucose will be determined in all samples, and a muscle biopsy will be collected post-prandially following the plant protein meal for examination of signalling markers of muscle plasticity (atrogin1, MURF1, LC3, BNIP3, Akt-dependent mTOR and FxO), metabolic adaptations (AMPK and PGC1alpha) and denervation (AChR subunits expression, agrin/MuSK/Lrp4, NCAM, and Myog) by UNIPD

ELIGIBILITY:
Inclusion Criteria:

* BMI 22-30 kg/m²
* Inactive (<150 minutes of moderate to vigorous physical activity per week and no regular resistance training),
* Covered by a social security system
* Agrees to undergo the study interventions (undirect calorimetry, functional tests, physical activity program)

Exclusion Criteria:

* Hamilton HAD scale with a score > 9
* Subject with a pathology or treatment (diabetic on insulin, corticosteroids > 8 days, neuroleptics, anticoagulant, antiplatelet) judged by the investigator as incompatible with the study
* Subject with unstabilized thyroid dysfunction for at least 3 months
* Subject with unstabilized hypertension for at least 3 months
* Subject with a medical and/or surgical history judged by the investigator as incompatible with the trial
* More than 21 alcoholic drinks per week
* Heavy smoker (>10 cigarettes/day)
* Currently participating in another intervention study
* Absence of informed consent
* Inability to participate in physical activity
* Allergy(ies) or refusal to consume one of the foods tested as part of the the study
* Allergy to local anesthetics
* Declared glaucoma
* Prostate hypertrophy
* Refusal to register in the national file of volunteers who participate in research involving human beings
* Subject in a period of exclusion from a previous study or having received a total amount of compensation greater than 6,000 euros over the 12 months preceding the start of the trial (after verification in the File of Volunteers for Research involving Human Beings)
* Patients under guardianship, curatorship, deprived of liberty or legal protection
* Subject with claustrophobia

Min Age: 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2025-08-26 (Actual); Primary Completion 2027-02 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
Splanchnic extraction of amino acids | At baseline (Week 0) and at follow-up (Weeks 12-13).
  Change in splanchnic extraction of amino acids in response to standardized test meals (vegetal & animal proteins), assessed before and after a 12-week physical activity program.

SECONDARY OUTCOMES:
Whole body protein metabolism | At baseline (Week 0) and at follow-up (Weeks 12-13).
  Evaluation of protein turnover and amino acid oxidation using peripheral blood samples and breath tests before and after a 12-week physical activity program.
Skeletal muscle signaling markers | At baseline (Week 0) and at follow-up (Weeks 12-13) following only the plant protein standardized meal
  Markers of plasticity, metabolism and denervation in skeletal muscle biopsy

CONTACTS AND LOCATIONS:
Overall Officials: Yves Boirie, Principal Investigator — CHU de Clermont-Ferrand
Locations (1):
- CHU de Clermont-Ferrand, Clermont-Ferrand, France

IPD SHARING:
Plan to Share IPD: Undecided